CLINICAL TRIAL: NCT05223725
Title: AdKCNH2-G628S Gene Therapy for Post-Operative Atrial Fibrillation
Brief Title: Gene Therapy for Post-Operative Atrial Fibrillation
Acronym: AFGT01
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Problems with receiving investigational agent and problems with funding
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: WIRB1333791
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Post-operative Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participant is masked due to delivery during general anesthesia, outcomes assessors and investigators are fully masked to study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- dose escalation (Experimental): initial phase, increasing dose
  Interventions: Biological: AdKCNH2-G628S
- low dose (Experimental): second phase, fixed dose 5x10(11) vp
  Interventions: Biological: AdKCNH2-G628S
- high dose (Experimental): second phase, fixed dose 2x10(12) vp
  Interventions: Biological: AdKCNH2-G628S
- control (No Intervention): second phase, blinded, randomized with no intervention delivered but with testing and monitoring.

INTERVENTIONS:
Biological: AdKCNH2-G628S — adenovirus containing the transgene KCNH2-G628S
  Arms: dose escalation; high dose; low dose

SUMMARY:
This clinical trial will have 2 components: a brief dose-ranging study and a randomized comparison of 2 doses of AdKCNH2-G628S with control cardiac surgery patients. The study will assess safety of the intervention in a population at increased risk for post-operative atrial fibrillation.

DETAILED DESCRIPTION:
Post-operative AF (POAF) is a specific form of AF occurring in the days after cardiothoracic surgery. A unique element of POAF is the limited duration of risk, which peaks 3 days and dissipates 10 days after surgery. We propose gene therapy for POAF. Our hypothesis is that counteracting AF-related electrical remodeling will disrupt the reentrant electrical circuits integral to maintaining AF. We have extensive preclinical data showing safety and efficacy of adenoviral gene transfer using the gene mutation KNCH2-G628S. When delivered to the atria using adenoviruses and a novel gene painting technique, KCNH2-G628S effectively and specifically prolongs atrial action potential and prevents development of AF for the 10-14-day duration of post-operative AF risk. This clinical trial will have 2 components: a brief dose-ranging study and a randomized comparison of 2 doses of AdKCNH2-G628S with control cardiac surgery patients.

ELIGIBILITY:
Inclusion:

* Elective valve surgery (alone or with coronary artery bypass grafting surgery) and one of the risk factors listed below, or elective coronary artery bypass grafting surgery with two of the risk factors listed below.
* Risk factors:

  * age greater than 70,
  * increased left atrial size (> 4 cm left atrial diameter or LA volume index > 35 on echocardiogram).
  * obesity (body mass index > 30)
  * history of:

    * paroxysmal AF
    * hypertension
    * chronic pulmonary disease
    * diabetes mellitus
    * clinical heart failure
    * rheumatic heart disease

Exclusion:

* persistent or permanent AF
* QTc > 475 on pre-op ECG or any time in last year (unless due to QT prolonging drug that was stopped > 5 half-lives before surgery with verification of QT normalization after discontinuing drug)
* QTc prolonging drug use (unless stopped > 5 half-lives prior to surgery)
* Any antiarrhythmic drug use in last year (inclusive of Vaughan Williams class I and III drugs, not including β-blocker or calcium channel blocker drugs)
* Any history of inherited arrhythmia syndrome
* Any prior or current sustained ventricular arrhythmias
* Any prior or current clinically significant bradyarrhythmias unless already treated with pacemaker and ventricular pacing <20% (to reliable measure QT interval during the study)
* Any prior gene therapy
* Left ventricular ejection fraction (LVEF) < 35%
* Prior open chest surgery
* History of or current malignancy, unless documented to be cured
* History of or current chemotherapy, radiotherapy, or other immunosuppressive therapy within the past 30 days. Corticosteroid treatment may be permitted at the discretion of the Primary Investigator
* History of infection with human immunodeficiency virus (HIV), hepatitis A, B, or C, or tuberculosis
* Immunizations of any kind in the month prior to surgery
* Underlying defect in immune function or history of multiple or severe life-threatening infections
* Significant liver disease (active hepatitis, AST or ALT greater than twice the upper limit of normal, prior or current liver failure with Pugh-Child category A-C disease)
* Significant renal disease (GFR less than 30)
* Current pregnancy
* Childbearing potential unless participant agrees to prevent pregnancy prior to and for at least 3 months after virus delivery 10
* Any condition that limits life to < 12 months other than the condition to be treated with the planned surgery
* Participation in any other clinical trial within 30 days of surgery
* Incarcerated persons
* Individuals under the age of 18 years
* Unwillingness to undergo the study interventions and follow-up as outlined in the schedule of events
* Ongoing medical or other condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study
* Lack of capacity to provide participant's own informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
proportion of patients having a post-operative complication relative to controls | 3 months
  proportion of patients having a post-operative complication relative to controls

SECONDARY OUTCOMES:
proportion of patients having post-operative atrial fibrillation | 1 month
  proportion of patients having post-operative atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Donahue, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMass Memorial Hospital, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the clinical trial will be made available to the scientific community and the general public in the following ways:
  1. As soon as final data are complete, verified and analyzed, manuscripts will be written and submitted to scientific journals with the highest possible impact factor to achieve the widest possible dissemination within the scientific community.
  2. Presentations at scientific meetings within the disciplines of cardiac surgery, cardiology, cardiac electrophysiology and gene therapy will further disseminate the research information gained as a result of the proposed studies.
  3. The research data will be uploaded to an openly available research website maintained by UMass for review and use by the scientific community.
  4. The research results will be uploaded to clinicaltrials.gov.
  5. Press releases, summaries of research findings and interviews with investigators will be released to the general public to publicize the information gained in the proposed research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: as per plan description
Access Criteria: as per plan description

REFERENCES:
- [Background] Kikuchi K, McDonald AD, Sasano T, Donahue JK. Targeted modification of atrial electrophysiology by homogeneous transmural atrial gene transfer. Circulation. 2005 Jan 25;111(3):264-70. doi: 10.1161/01.CIR.0000153338.47507.83. Epub 2005 Jan 10. PMID 15642761
- [Background] Amit G, Kikuchi K, Greener ID, Yang L, Novack V, Donahue JK. Selective molecular potassium channel blockade prevents atrial fibrillation. Circulation. 2010 Jun 1;121(21):2263-70. doi: 10.1161/CIRCULATIONAHA.109.911156. Epub 2010 May 17. PMID 20479154
- [Background] Liu Z, Hutt JA, Rajeshkumar B, Azuma Y, Duan KL, Donahue JK. Preclinical efficacy and safety of KCNH2-G628S gene therapy for postoperative atrial fibrillation. J Thorac Cardiovasc Surg. 2017 Nov;154(5):1644-1651.e8. doi: 10.1016/j.jtcvs.2017.05.052. Epub 2017 May 23. PMID 28676183